CLINICAL TRIAL: NCT05886010
Title: Evaluation of the Performance and Tolerance of Cyto-selective Difluoroethane-based Cryotherapy in th Treatment of Brown Spots (Solar and Senile Lentigines, Post-Inflammatory Hyperpigmentation) on the Face and Hands of Asian Ethnicity Skins
Brief Title: Performance and Tolerance of Cyto-selective Difluoroethane-based Cryotherapy in th Treatment of Brown Spots (Solar and Senile Lentigines, Post-Inflammatory Hyperpigmentation) on the Face and Hands of Asian Ethnicity Skins
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cryonove Pharma (Industry)
Collaborators: CEISO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CS5_4
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Solar Lentigo; Senile Lentigo
Keywords: Cryotherapy; Hyperpigmentation; Skin Diseases
MeSH Terms: conditions — Hyperpigmentation; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Condition 1 :prototypes 1 everyday (Experimental): Application on the brown spots of the face and the hands for the prototypes 1 at D0,D1,D2,D3,D4 and D5
  Interventions: Device: prototypes 1 everyday
- Condition 2 : prototypes 1 every week (Experimental): Application on the brown spots of the face and the hands for the prototypes 1 at D0,D7,D14,D21,D28, D35, D42, D49, D56, D63, D70 and D77.
  Interventions: Device: prototypes 1 every week
- Condition 3 : prototypes 1 every two weeks (Experimental): Application on the brown spots of the face and the hands for the prototypes 1 at D0,D14,D28, D42, D56 and D70
  Interventions: Device: prototypes 1 every two weeks
- Condition 4 : prototypes 2 every two weeks (Experimental): Application on the brown spots of the face and the hands for the prototypes 2 at D0,D14,D28, D42, D56 and D70
  Interventions: Device: prototypes 2 every two weeks
- Condition 5 : prototypes 3 every two weeks (Experimental): Application on the brown spots of the face and the hands for the prototypes 3 at D0,D14,D28, D42, D56 and D70
  Interventions: Device: prototypes 3 every two weeks

INTERVENTIONS:
Device: prototypes 1 everyday — Application on brown spots located on the face and/or the hand (6 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face or/and hand. Subjects will be lying down, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 1 :prototypes 1 everyday
Device: prototypes 1 every week — Application on brown spots located on the face and/or the hand (12 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face or/and hand. Subjects will be lying down, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 2 : prototypes 1 every week
Device: prototypes 1 every two weeks — Application on brown spots located on the face and/or the hand (6 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face or/and hand. Subjects will be lying down, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 3 : prototypes 1 every two weeks
Device: prototypes 2 every two weeks — Application on brown spots located on the face and/or the hand (6 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face or/and hand. Subjects will be lying down, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 4 : prototypes 2 every two weeks
Device: prototypes 3 every two weeks — Application on brown spots located on the face and/or the hand (6 treatments during the study). An operator previously trained by the dermatologist will apply the study device to the patient's face or/and hand. Subjects will be lying down, and the prototypes will be administered upside down for the applications on the face and sitting for the applications on the hands. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas.
  Arms: Condition 5 : prototypes 3 every two weeks

SUMMARY:
CS5_4 study aim to evaluate the performance and the tolerance of 3 prototypes of cyto-selective cryotherapy treatments applied on the brown spots on the face and hands of asian ethnicity skins (chinese). A brown spot is defined as solar or senile lentigo (SSL) and post-inflammatory hyperpigmentation (PIH).

Each treatment corresponds to a combination of a specific sequence of cryogenic spray and of a frequency of application. Each spot will be treated by a defined prototype (always the same device on the same spot all along the study).

The study will evaluate the following prototype :

* Prototypes 1
* Prototypes 2
* Prototypes 3

DETAILED DESCRIPTION:
Rational :

Solar/senile lentigo (SSL) is a harmless patch of darkened skin. It results from exposure to ultraviolet (UV) radiation, which causes local proliferation of melanocytes and accumulation of melanin within the skin cells (keratinocytes). Solar/senile lentigos or lentigines are very common, especially in people over the age of 40 years. Solar/senile lentigines are found as groups of similar lesions on sun-exposed sites, particularly the face or the back of hands.

Post-inflammatory hyperpigmentation (PIH) is an area of darker skin that remains after a pimple or wound heals. The discoloration is due to the production of excess melanin (pigment) as part of the skin's natural response to inflammation.

CRYONOVE is a medical device intended to induce a cyto-selective cryogenic action on melanocytes to remove brown spots resulting from solar or senile lentigines, post-inflammatory hyperpigmentation and melasma on the face and body.

Cryotherapy is more and more used to improve skin appearance and currently used to treat lentigo spot. Devices using difluoroethane, manufactured by CRYONOVE PHARMA, are already available on the local and international markets, e.g. CRYOBEAUTY MAINS and CRYOBEAUTY CORPS.

However, the cryogenic gas (conventional cryotherapy - liquid nitrogen) creates a dermabrasion of the skin surface and person receiving this kind of treatment presents an impaired skin during a few days following the treatment as temporary damage of stratum corneum, erythema, scars, burns.

Following the side effects occurring after conventional cryotherapy application, it seems interesting for the sponsor to select other sequences of a cryogenic spray (3 prototypes of devices for face and hands used according to different frequencies of application, i.e., 5 conditions evaluated) which could be used for lentigo and post inflammatory hyperpigmentation treatment in Asian Ethnicity Skin with a same benefit for the consumers without any safety outcomes.

Design:

The study performed is a proof of concept, exploratory, interventional, monocentric, randomized and single blinded

Intervention :

3 prototypes of devices are evaluated in 5 different conditions. Each treatment corresponds to a combination of a specific sequence of cryogenic spray and of a frequency of application.

For the conditions 1, 3, 4 and 5, each spot will be treated 6 times during the study :

* Every day from D0 and thus until D5 (condition 1);
* Every two weeks: at D0, D14, D28, D42, D56 and at D70 (condition 3):
* Every two weeks: at D0, D14, D28, D42, D56 and at D70 (condition 4);
* Every two weeks: at D0, D14, D28, D42, D56 and at D70 (condition 5).

For the condition 2, each spot will be treated 12 times during the study:

• Every week: at D0, D7, D14, D21, D28, D35, D42, D49, D56, D63, D70 and at D77 (condition 2);

120 participant will be included in the study. Overall, this study leads to treat 240 face spots (PIH, SSL) and 40 hands spots (SSL) with 3 prototypes having different temperature and kinetic.

Prior to any study device application, the dermatologist will assess the adverse events and will decide if the period between two consecutive applications should be extended or not.The dermatologist will verify that the skin has not been treated by cosmetic products (no presence of cream that could interfere with the treatment) and is dry.

An operator previously trained by the dermatologist will apply the study device to the patient's face or hands. Subjects will be lying down, and the device will be administered upside down. During applications on the face, subjects will wear diving goggles protecting the eyes from cryogenic gas. For the application on the hands, the hands will be placed flat on the table and the prototypes will be applied upside down.The treatment will be stoped after the disappearance of the spot.

The patient follow-up visits are from Day 0 to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female or male,
* Chinese ethnicity skins,
* Ages between 18 years old and 75 years old,
* Phototype II or III (according to Fitzpatrick scale),
* Featuring brown spots ≥ 3 and ≤ 6 mm in diameter
* Agreeing not to be exposed to the sun (or artificial UV) during the study.
* Informed, having undergone a general clinical examination attesting to his/her ability to participate in the study.
* Having given written consent for their participation in the study.
* No suspicion of carcinoma after investigation by a dermatologist.

Exclusion Criteria:

* Having performed cosmetic treatments (exfoliants, scrubs or self-tanners, manicures, facials, UV ...) in the month before the start of the study where the prototypes will be applied.
* Having applied a depraving product in the month prior to the start of the study, where the prototypes will be applied.
* Having performed cosmetic treatments in a dermatologist (laser, Intense Pulsed Light (IPL), peeling, creams, cryotherapy ...) in the last 6 months where the prototypes will be applied (see restrictions paragraph).
* With dermatosis, autoimmune disease, systemic, chronic or acute disease, or any other pathology that may interfere with treatment or influence the results of the study (people with diabetes or circulatory problems, allergic to cold, Raynaud's syndrome...).
* Receiving treatment by general or local (dermo corticoids, corticosteroids, diuretics ...) Likely to interfere with the evaluation of the parameter studied.
* Participating in another study or being excluded from a previous study.
* Unable to follow the requirements of the protocol.
* Vulnerable: whose ability or freedom to give or refuse consent is limited.
* Major protected by law (tutorship, curatorship, safeguarding justice...).
* People unable to read and write the language of the documents involved in the study.
* Unable to be contacted urgently over the phone.

For female subjects:

* Pregnant woman (or wishing to be pregnant during study) or while breastfeeding.
* A woman who does not have a contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Change from baseline skin hyperpigmentation | Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, Day 91, Day 0 + 6 months
  The evaluation will be performed visually on the selected spots.
  A scale in 6 points (0 to 5) will be used :
  0=Clear of hyperpigmentation;
  1. Almost clear of hyperpigmentation;
  2. mild, but noticeable hyperpigmentation;
  3. moderate hyperpigmentation (medium brown in quality);
  4. severe hyperpigmentation (dark brown in quality);
  5. very severe hyperpigmentation (very dark brown, almost black in quality).
Change from baseline skin hypopigmentation | Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, Day 91, Day 0 + 6 months
  The evaluation will be performed visually on the selected spots.
  A scale in 5 points will be used (0 to 4):
  0=no hypopigmented lesion;
  1. very slight area of hypopigmentation of very small size and very slightly fairer than the surrounding skin;
  2. slight area of hypopigmentation of small size and slightly fairer than the surrounding skin;
  3. moderate : area of hypopigmentation of moderate size and much fairer than the surrounding skin;
  4. severe : area of hypopigmentation of large size and much fairer than the surrounding skin.
Change from baseline skin appearance - expected events | Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, Day 91, Day 0 + 6 months
  The evaluation will be performed visually on the selected spots and surrounded spotless skin area around the spot skin to assess erythema, oedema blister, bubble, scars, micro-bruise, hematoma, dryness,desquamation, fissures/cracks, roughness,crust, pink spots and papules.
  A scale in 5 points (0 to 4) will be used :
  0=none;
  1. very mild;
  2. mild;
  3. moderate;
  4. severe.
Change from baseline skin sensation | Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, Day 91, Day 0 + 6 months
  The evaluation will be performed visually on the selected spots and around the spot skin to assess tightness, stinging, itching, warm and burning sensation.
  A scale in 5 points (0 to 4) will be used :
  0=none;
  1. very mild;
  2. mild;
  3. moderate;
  4. severe.
Self-assesment of pain by VAS | Day 0
  The pain of the treatment will be assessed by the Visual Analogue Scale (VAS) at time T0 on the treated area.
  The pain assessed is that felt during the application of the devices. It will be collected from the patient within 5 minutes of application. The VAS is made up of a 10-centimeter line anchored by two ends of the pain. 10 is the first end being the "maximum pain imaginable" and 0 is the other end being "no pain".
Change from baseline spots visibility | Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 49, Day 56, Day 63, Day 70, Day 77, Day 91, Day 0 + 6 months
  Standardized photographs will be taken using a Dermatoscope C-Cube® (PIXIENCE) which allows realizing high resolution skin pictures. The capture will be taken on the previously selected lentigo and a spotless area.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Cadot, Principal Investigator — Laboratoir BIO-EC
Locations (1):
- Laboratoire BIO-EC, Longjumeau, France